CLINICAL TRIAL: NCT02867618
Title: Phase I/II Study of Carfilzomib and a PI3Kdelta Inhibitor TGR-1202 in the Treatment of Patients With Relapsed or Refractory Lymphoma
Brief Title: Carfilzomib and TGR-1202 in Treatment of R/R Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAP5661
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Hodgkin Disease; Lymphoma, Non-hodgkin
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — carfilzomib; umbralisib; rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carfilzomib + TGR-1202 (Experimental): Oral TGR-1202 will be given PO once daily on Days 1-28 and carfilzomib given intravenously twice a week for 3 consecutive weeks, on days 1, 2, 8, 9, 15, and 16 on the 28-day cycle.
  Interventions: Drug: Carfilzomib; Drug: TGR-1202

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib given intravenously twice a week for 3 consecutive weeks, on days 1, 2, 8, 9, 15, and 16 on the 28-day cycle. This will be in combination with the oral TGR-1202
  Other Names: Kyprolis
Drug: TGR-1202 — Oral TGR-1202 will be given PO once daily on Days 1-28 . This will be given in combination with the intravenous Carfilzomib
  Other Names: (formerly) RP-5264

SUMMARY:
This is an open label, phase I/II, dose-escalation study in the initial phase I followed by a phase II.

The primary objective of the phase I is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of the combinations of TGR-1202 and carfilzomib in participants with relapsed and refractory (R/R) non-Hodgkin lymphoma (NHL) and Hodgkin lymphoma (HL). The safety and toxicity of this combination will be evaluated throughout the entire study.

If the combination of TGR-1202 and carfilzomib is found to be feasible and an MTD is established, the phase II part of the study will be initiated.

Phase II will consist of a 2-stage design of the combination of TGR-1202 and carfilzomib for participants with R/R NHL.

DETAILED DESCRIPTION:
Dysregulated c-Myc is associated with resistance to chemotherapy and poor survival in aggressive lymphomas. Novel strategies that target this biology could markedly improve the outcome of these participants. To date no drugs that directly target Myc have been approved for cancer treatment. Recent results by Deng et al. (Blood. 2017 Jan 5. PMID: 27784673) described a highly synergistic regimen discovered in preclinical models, through combining TGR-1202, an investigational drug that inhibits PI3K delta, and carfilzomib, a drug approved by the FDA for multiple myeloma. Importantly, the combination of TGR-1202 and carfilzomib acts by potently silencing the translation of c-Myc and inducing apoptosis in many cell lines and primary lymphoma cells representing broad histological subtypes of lymphoma. These results suggest that TGR-1202 and carfilzomib may be highly effective in relapsed and refractory lymphoma where c-Myc plays a key pathological role.

ELIGIBILITY:
Target Population Phase I: Patients with relapsed or refractory NHL and HL Phase II: Patients with relapsed or refractory NHL

Inclusion Criteria:

* Phase I: Patients must have histologically confirmed R/R NHL or HL (defined by World Health Organization (WHO) criteria). Patients with chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL) are eligible. In addition, patients with NHL other than diffuse large B cell lymphomas (DLBCL) must have received at least 2 prior therapies. Patients with DLBCL and HL will be eligible if there is no available standard therapy.
* Phase II: Patients must have histologically confirmed R/R NHL (as defined by WHO criteria). Patients with NHL other than diffuse large B cell lymphomas (DLBCL) must have received at least 2 prior therapies. Patients with DLBCL will be eligible if there is no available standard therapy.
* Must have received front line chemotherapy. No upper limit for the number of prior therapies
* Evaluable Disease in the Phase I, and measurable disease in the Phase II
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Patients must have adequate organ and marrow function
* Adequate Contraception
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Prior Therapy Exposure to chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier. Systemic steroids that have not been stabilized (≥ 5 days) to the equivalent of ≤10 mg/day prednisone prior to the start of the study drugs. No other investigational agents are allowed.
2. History of allergic reactions to TGR-1202 or carfilzomib
3. Uncontrolled inter-current illness
4. Pregnant women
5. Nursing women
6. Current malignancy or history of a prior malignancy
7. Patient known to be Human Immunodeficiency Virus (HIV)-positive
8. Active Hepatitis A, Hepatitis B, or Hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Changchun Deng, MD, Principal Investigator — Assistant Professor of Clinical Medicine and Experimental Therapeutics
Locations (1):
- Columbia University Irving Medical Center - Center for Lymphoid Malignancies, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 out of 14 subjects were enrolled (consented) but not accrued into study and did not receive study treatment.
Period: Overall Study
Arm/Group | Carfilzomib + TGR-1202
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 3 out of 14 subjects were enrolled but not accrued into study; however, baseline information was collected for all 14 subjects.
Arm/Group | Carfilzomib + TGR-1202
Number analyzed (Participants) | 14
Age, Customized [Number; unit: participants]
  18-21 years | 0
  22-29 years | 1
  30-39 years | 1
  40-49 years | 0
  50-59 years | 1
  60-69 years | 2
  70-79 years | 9
  80-89 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase 1) - TGR-1202 Only
Description: The highest dose of the study treatment that does not cause unacceptable side effects.
Time Frame: 9 months
Population: PI left the institution, study data was not complete or analyzed for Carfilzomib (Phase 2).
Measure: Number; unit: mg
Arm/Group | Carfilzomib + TGR-1202
Number analyzed (Participants) | 11
mg | 800

2. Primary Outcome: Objective Response Rate (ORR) (Phase 2)
Description: Defined as best response (complete response and partial response) by 4 cycles.
Time Frame: 9 months
Population: The data was not collected or analyzed due to PI leaving the institution.
Arm/Group | Carfilzomib + TGR-1202
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year post study treatment
Arm/Group | Carfilzomib + TGR-1202
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib + TGR-1202 (N=11)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Grade 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT02867618/Prot_SAP_000.pdf